CLINICAL TRIAL: NCT06503016
Title: The Effect of phoSPHocreatine on mEdical Emergency Team (Met) tREated Patients: a Randomized Clinical Trial Protocol
Brief Title: The Effect of phoSPHocreatine on mEdical Emergency Team (Met) tREated Patients
Acronym: SPHERE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Collaborators: Silvia Ajello (Unknown)
Responsible Party: Principal Investigator, Giovanni Landoni, MD, Full Professor, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GR-2021-12375001
Record Dates: First submitted 2024-07-05; First posted 2024-07-16 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Hypotension; Consciousness, Level Altered; Airway Disease; Respiratory Failure; Tachypnea; Bradypnea; Tachycardia; Bradycardia; Cardiac Failure; Cardiac Arrest
MeSH Terms: conditions — Hypotension; Consciousness Disorders; Respiratory Insufficiency; Tachypnea; Hypoventilation; Tachycardia; Bradycardia; Heart Failure; Heart Arrest | interventions — Phosphocreatine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phosphocreatine (Experimental): Patients randomized to the phosphocreatine group will receive the drug for a maximum of 3 days.
  * Patients without renal failure: At the time of randomization (day 0), 4 grams of phosphocreatine will be administered, followed by an additional 4 grams on the same day, with a minimum interval of 20 minutes and a maximum of 4 hours. On day 1 and day 2, after 8 AM, 2 grams of phosphocreatine will be administered twice a day, with a 6-hour interval between doses.
  * Patients with history of renal failure: On day 0, patients will receive a single dose of 4 grams of phosphocreatine. On day 1 and day 2, after 8 AM, 2 grams of phosphocreatine will be administered twice a day, with a 6-hour interval between doses.
  * Patients with acute kidney injury, without chronic kidney disease: Single dose of 4 grams of phosphocreatine on day 0. No further doses of the drug are planned.
  Interventions: Drug: Phosphocreatine
- Placebo (Placebo Comparator): Patients randomized to the placebo group will receive saline solution for a maximum of 3 days.
  * Patients without renal failure: 200 ml of saline solution twice a day from day 0 to day 2. On day 0, the second bolus should be administered between 20 minutes and 4 hours after the first bolus; on day 1 and day 2, the saline solution should be administered after 8 AM, with the second bolus given 6 hours later.
  * Patients with history of renal failure: On day 0, a single infusion of 200 mL of saline solution will be administered. On day 1 and day 2, 200 mL of saline solution will be administered twice a day, after 8 AM, with a 6-hour interval between doses.
  * Patients with acute kidney injury, without chronic kidney disease: A single infusion of 200 mL of saline solution on day 0. No further administrations are planned.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Phosphocreatine — Administration of Phosphocreatine
  Arms: Phosphocreatine
Drug: Placebo — Saline solution of NaCl 0.9%
  Arms: Placebo

SUMMARY:
Unexpected deaths and unplanned intensive care unit (ICU) admissions are common during hospital stay and are often preceded by warning abnormalities in patients' vital signs. These abnormalities trigger Medical Emergency Team (MET) activation and up to 15% of patients visited by the MET is admitted to the ICU with an overall hospital stay after the MET intervention of approximately 2 weeks. Phosphocreatine (PCr) is a natural energy-buffering molecule associated with signals of mortality reduction in patients with acute cardiac conditions (according to meta-analytic finding from our group) and with encouraging beneficial effects on other acute organ failures (e.g. brain). The investigators designed a multi-center, randomized, placebo-controlled trial to confirm the promising beneficial effects of PCr in hospitalized patients. The investigators expects a reduction in hospital stay (measured as an increase in days alive and out of hospital at 30 days) when PCr is added to standard treatment in patients requiring MET intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted in hospital (but outside ICU)
2. Age>=18 years
3. Written informed consent
4. Serum creatinine <=2 mg/dl
5. Patient with impending or underlying cardiac failure or cardiac arrest, irrespectively of the primitive organ failure, and the Medical Emergency Team (MET) is called upon at least one of the following:

   1. Threatened airways;
   2. Respiratory arrest;
   3. Respiratory rate <5 or >36 breaths per min;
   4. Pulse rate <40 or >140 beats per min;
   5. Systolic blood pressure < 90 mm Hg;
   6. Sudden fall in level of consciousness;
   7. Fall in Glasgow coma scale of > 2 points.

Exclusion Criteria:

1. Age < 18 years;
2. Ongoing cardiac massage;
3. Current hospital admission from a care nursing facility;
4. Planned discharge to a care nursing facility;
5. Reasons for withdrawal of life-sustaining therapy;
6. History of kidney transplantation;
7. Solitary kidney (by any reason);
8. Serum Creatinine > 2 mg/dl;
9. Immediate need for ICU admission;
10. Known allergy to PCr;
11. Pregnancy;
12. Previous enrollment and randomization into this trial;
13. Administration of PCr in the previous 30 day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
days alive and out of hospital at 30 days. | day 30 or hospital discharge
  To compare the effect of phosphocreatine (PCr) (experimental group), versus placebo (saline solution-control group) on the number of days alive and out of hospital at 30 days.

SECONDARY OUTCOMES:
Cognitive function | day 30
  Evaluation of cognitive function using the Cognitive Telephone Screening Instrument (COGTEL). The COGTEL is a test that evaluates the cognitive performance of survived patients 30 days after randomization. This scale has a minimum of zero points and a maximum of 100.
Rate of arrhythmia needing treatment | hospital discharge (which usually occurs in the 30days after randomization)
  Clinically relevant arrhythmias will be recorded and confirmed by an ECG. Rate of major arrhythmias divided into supraventricular arrhythmias, ventricular arrhythmias, bradyarrhythmias, and need for antiarrhythmics will be registered.
Rate of ICU admissions or criteria for ICU admission | hospital discharge (which usually occurs in the 30days after randomization)
  ICU admission
Death at 30 days | day 30
  Death
Death at 90 days | 90 days
  Death

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, Italy

REFERENCES:
- [Background] Landoni G, Zangrillo A, Lomivorotov VV, Likhvantsev V, Ma J, De Simone F, Fominskiy E. Cardiac protection with phosphocreatine: a meta-analysis. Interact Cardiovasc Thorac Surg. 2016 Oct;23(4):637-46. doi: 10.1093/icvts/ivw171. Epub 2016 Jun 17. PMID 27318357
- [Background] Mingxing F, Landoni G, Zangrillo A, Monaco F, Lomivorotov VV, Hui C, Novikov M, Nepomniashchikh V, Fominskiy E. Phosphocreatine in Cardiac Surgery Patients: A Meta-Analysis of Randomized Controlled Trials. J Cardiothorac Vasc Anesth. 2018 Apr;32(2):762-770. doi: 10.1053/j.jvca.2017.07.024. Epub 2017 Jul 24. PMID 29409711